CLINICAL TRIAL: NCT01196416
Title: Phase Ib/II Study of the Gamma-Secretase Inhibitor (GSI) RO4929097 in Combination With Cisplatin, Vinblastine, and Temozolomide (CVT) in Patients With Metastatic Melanoma
Brief Title: Gamma-secretase/Notch Signalling Pathway Inhibitor RO4929097 in Combination With Cisplatin, Vinblastine, and Temozolomide in Treating Patients With Recurrent or Metastatic Melanoma
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2011-02524; NCI-2011-02524 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000684220; 10-085 (Other: Memorial Sloan-Kettering Cancer Center); 8491 (Other: CTEP); N01CM62206 (NIH); P30CA008748 (NIH); U01CA069856 (NIH)
Record Dates: First submitted 2010-09-04; First posted 2010-09-08 (Estimated); Results first posted 2017-10-18 (Actual); Last update posted 2019-11-18 (Actual); Status verified 2019-10

CONDITIONS: Recurrent Melanoma; Stage IV Skin Melanoma
MeSH Terms: conditions — Melanoma | interventions — Cisplatin; 1,2-diaminocyclohexaneplatinum II citrate; Platinum; 2,2-dimethyl-N-(6-oxo-6,7-dihydro-5H-dibenzo(b,d)azepin-7-yl)-N'-(2,2,3,3,3-pentafluoropropyl)malonamide; Temozolomide; Vinblastine

ARMS (1):
- Treatment (RO4929097, cisplatin, vinblastine, temozolomide) (Experimental): Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO QD on days 1-21, cisplatin IV over 30 minutes and vinblastine IV over 30 minutes on days 1-3, and temozolomide PO QD on days 1-5. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients without progressive disease continue to receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 and temozolomide as above in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Cisplatin; Drug: Gamma-Secretase Inhibitor RO4929097; Other: Laboratory Biomarker Analysis; Other: Pharmacological Study; Drug: Temozolomide; Drug: Vinblastine Sulfate

INTERVENTIONS:
Drug: Cisplatin — Given IV
  Other Names: Abiplatin; Blastolem; Briplatin; CDDP; Cis-diammine-dichloroplatinum; Cis-diamminedichloridoplatinum; Cis-diamminedichloro Platinum (II); Cis-diamminedichloroplatinum; Cis-dichloroammine Platinum (II); Cis-platinous Diamine Dichloride; Cis-platinum; Cis-platinum II; Cis-platinum II Diamine Dichloride; Cismaplat; Cisplatina; Cisplatinum; Cisplatyl; Citoplatino; Citosin; Cysplatyna; DDP; Lederplatin; Metaplatin; Neoplatin; Peyrone's Chloride; Peyrone's Salt; Placis; Plastistil; Platamine; Platiblastin; Platiblastin-S; Platinex; Platinol; Platinol- AQ; Platinol-AQ; Platinol-AQ VHA Plus; Platinoxan; Platinum; Platinum Diamminodichloride; Platiran; Platistin; Platosin
Drug: Gamma-Secretase Inhibitor RO4929097 — Given PO
  Other Names: RO4929097
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Pharmacological Study — Correlative studies
Drug: Temozolomide — Given PO
  Other Names: CCRG-81045; Imidazo[5,1-d]-1,2,3,5-tetrazine-8-carboxamide, 3, 4-dihydro-3-methyl-4-oxo-; M & B 39831; M and B 39831; Methazolastone; RP-46161; SCH 52365; Temodal; Temodar
Drug: Vinblastine Sulfate — Given IV
  Other Names: 29060 LE; 29060-LE; Exal; Velban; Velbe; Velsar; VINCALEUKOBLASTINE

SUMMARY:
This phase Ib/II trial studies the side effects and best dose of gamma-secretase/Notch signalling pathway inhibitor RO4929097 when given together with cisplatin, vinblastine, and temozolomide and to see how well they work in treating patients with recurrent or metastatic melanoma. Gamma-secretase/Notch signalling pathway inhibitor RO4929097 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Drugs used in chemotherapy, such as cisplatin, vinblastine, and temozolomide, work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving gamma-secretase/Notch signalling pathway inhibitor RO4929097 together with combination chemotherapy may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To characterize the safety and tolerability of daily RO4929097 (gamma-secretase/Notch signalling pathway inhibitor RO4929097) administered orally daily in combination with CVT (starting dose: cisplatin 25 mg/m^2 intravenous [IV] daily x 3; vinblastine 1.2 mg/m^2 IV daily x 3, and temozolomide [TMZ] 150 mg/m^2 orally [PO] daily x 5) administered on an every 21 day schedule. (Phase Ib) II. To determine the maximum-tolerated dose (MTD) of RO4929097 with CVT in patients with metastatic melanoma with correlative biomarkers for Notch pathway signaling and gamma secretase enzyme activity. (Phase Ib) III. Based on the MTD from the phase Ib study, to conduct a phase II trial and to determine the response rate and overall survival. (Phase II)

SECONDARY OBJECTIVES:

I. To describe the pharmacokinetics and pharmacodynamics of the combination of RO4929097 and temozolomide. (Phase Ib) II. To obtain tissue biopsy for correlative studies before the initiation of therapy and one week after treatment with RO4929097 and CVT. (Phase Ib and II) III. To determine the progression-free survival of patients treated at the phase II dose. (Phase II)

OUTLINE: This is phase I dose-escalation study of gamma-secretase inhibitor RO4929097, followed by a phase II study.

Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 PO once daily (QD) on days 1-21, cisplatin IV over 30 minutes and vinblastine IV over 30 minutes on days 1-3, and temozolomide PO QD on days 1-5. Treatment repeats every 21 days for 6 courses in the absence of disease progression or unacceptable toxicity. Patients without progressive disease continue to receive gamma-secretase/Notch signalling pathway inhibitor RO4929097 and temozolomide as above in the absence of disease progression or unacceptable toxicity.

After completion of study therapy, patients are followed up for 24 months.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically or cytologically Memorial Sloan Kettering Cancer Center (MSKCC) confirmed recurrent or metastatic melanoma
* All Patients must have measurable disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1; measurable disease is defined as at least one lesion that can be accurately measured in at least one dimension (longest diameter to be recorded); each lesion must be > 10 mm when measured by computed tomography (CT), magnetic resonance imaging (MRI) or caliper measurement by clinical exam; or > 20 mm when measured by chest x-ray; lymph nodes must be > 15 mm in short axis when measured by CT or MRI
* Patients may have had up to one prior systemic therapy for recurrent or metastatic disease, but cannot have previously been treated with cisplatin, vinblastine, temozolomide, dacarbazine, or a gamma-secretase inhibitor; at least 3 weeks must have elapsed since the last dose of systemic therapy; for small molecule targeted therapy, at least 5 half-lives must have elapsed; at least 6 weeks must have elapsed if the last regimen included carmustine (BCNU) or mitomycin C or an anti-cytotoxic T-lymphocyte antigen 4 (CTLA4) antibody
* Life expectancy of greater than 3 months
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2 (Karnofsky >= 60%)
* Hemoglobin >= 9 g/dL
* Leukocytes >= 3,000/mcL
* Absolute neutrophil count >= 1,500/mcL
* Platelets >= 100,000/mcL
* Total bilirubin =< institutional upper limit of normal
* Aspartate aminotransferase (AST) (serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 X institutional upper limit of normal
* Creatinine within normal institutional limits OR creatinine clearance >= 60 mL/min/1.73 m^2 for patients with creatinine levels above institutional normal
* Women of childbearing potential and men must use two forms of contraception (i.e., barrier contraception and one other method of contraception) at least 4 weeks prior to study entry, for the duration of study participation, and for at least 12 months post-treatment; should a woman become pregnant or suspect she is pregnant while she or her partner are participating in this study and for 12 months after study participation, the patient should inform the treating physician immediately
* Women of childbearing potential are required to have a negative serum pregnancy test (with a sensitivity of at least 25 mIU/mL) within 10-14 days and within 24 hours prior to the first dose of RO4929097 (serum or urine); a pregnancy test (serum or urine) will be administered every 4 weeks if their menstrual cycles are regular or every 2 weeks if their cycles are irregular while on study within the 24-hour period prior to the administration of RO4929097; a positive urine test must be confirmed by a serum pregnancy test; prior to dispensing RO4929097, the investigator must confirm and document the patient's use of two contraceptive methods, dates of negative pregnancy test, and confirm the patient's understanding of the teratogenic potential of RO4929097
* Female patients of childbearing potential are defined as follows:

  * Patients with regular menses
  * Patients, after menarche with amenorrhea, irregular cycles, or using a contraceptive method that precludes withdrawal bleeding
  * Women who have had tubal ligation
* Female patients may be considered to NOT be of childbearing potential for the following reasons:

  * The patient has undergone total abdominal hysterectomy with bilateral salpingo-oophorectomy or bilateral oophorectomy
  * The patient is medically confirmed to be menopausal (no menstrual period) for 24 consecutive month
  * Pre-pubertal females; the parent or guardian of young female patients who have not yet started menstruation should verify that menstruation has not begun; if a young female patient reaches menarche during the study, then she is to be considered as a woman of childbearing potential from that time forward
* Ability to understand and the willingness to sign a written informed consent document
* Patients with accessible tumor must agree to undergo pre- and post-treatment tumor biopsies

Exclusion Criteria:

* Patients who have had chemotherapy or radiotherapy within 3 weeks (6 weeks for nitrosoureas or mitomycin C) prior to entering the study or those who have not recovered from adverse events due to agents administered more than 3 weeks earlier
* Patients may not be receiving any other investigational agents
* Patients with known brain metastases are excluded unless brain metastases have been resected or successfully treated with stereotactic radiosurgery and the patient has been free from central nervous system (CNS) recurrence or progression for 3 months
* History of allergic reactions attributed to compounds of similar chemical or biologic composition to RO4929097 or other agents used in the study
* Patients taking medications with narrow therapeutic indices that are metabolized by cytochrome P450 (CYP450), including warfarin sodium (Coumadin®) are ineligible
* Preclinical studies indicate that RO4929097 is a substrate of CYP3A4 and inducer of CYP3A4 enzyme activity; caution should be exercised when dosing RO4929097 concurrently with CYP3A4 substrates, inducers, and/or inhibitors; furthermore, patients who are taking concurrent medications that are strong inducers/inhibitors or substrates of CYP3A4 should be switched to alternative medications to minimize any potential risk; the following medications with strong potential for interaction are not allowed: indinavir, nelfinavir, ritonavir, clarithromycin, itraconazole, ketoconazole, nefazodone
* Patients with malabsorption syndrome or other condition that would interfere with intestinal absorption
* Patients must be able to swallow tablets
* Patients who are serologically positive for hepatitis A, B or C, and have an active infection, or have a history of liver disease, other forms of hepatitis or cirrhosis are ineligible
* Patients with uncontrolled electrolyte abnormalities including hypocalcemia, hypomagnesemia, hyponatremia, hypophosphatemia or hypokalemia, defined as less than the lower limit of normal for the institution, despite adequate electrolyte supplementation are excluded from this study
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, a history of torsades de pointes or other significant cardiac arrhythmias other than chronic, stable atrial fibrillation that require antiarrhythmics or other medications known to prolong corrected QT interval (QTc); psychiatric illness/social situations that would limit compliance with study requirements; patients may have had another cancer but there must be convincing clinical evidence that the melanoma is the disease requiring therapeutic intervention
* Pregnant women are excluded from this study; breastfeeding should be discontinued if the mother is treated with RO4929097; these potential risks may also apply to other agents used in this study
* HIV-positive patients on combination antiretroviral therapy are ineligible; appropriate studies will be undertaken in patients receiving combination antiretroviral therapy when indicated
* Cardiovascular: baseline QTc > 450 msec (male) or QTc > 470 msec (female)
* Patients who have not recovered to < Common Terminology Criteria for Adverse Events (CTCAE) grade 2 toxicities related to prior therapy are not eligible to participate in this study

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2010-08; Primary Completion 2015-08 (Actual); Study Completion 2015-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Mark Dickson, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (1):
- Memorial Sloan-Kettering Cancer Center, New York, New York, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide): Patients receive gamma-secretase/Notch signalling pathway inhibitor RO4929097, vinblastine and temozolomide
Period: Overall Study
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Started | 14
Completed | 12
Not Completed | 2
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Number analyzed (Participants) | 14
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 7
  >=65 years | 7
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 7

OUTCOME MEASURES:

1. Primary Outcome: Overall Objective Response
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progression, as a 20% increase in the sum of the longest diameter of target lesions, or a measurable increase in a non-target lesion, or the appearance of new lesions; Stable Disease (SD), neither sufficient shrinkage to qualify for PR nor sufficient increase to qualify for disease progression
Time Frame: From the time measurement criteria are met for CR or PR until the first date that recurrent or progressive disease is objectively documented, assessed up to 2 years
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Number analyzed (Participants) | 12
Participants
  Partial Response (PR) | 3
  Stable Disease (SD) | 3
  Progression of Disease (POD) | 6

2. Primary Outcome: Maximum-tolerated Dose for Cisplatin, Vinblastine and TMZ
Description: based on the incidence of dose-limiting toxicity as assessed the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase IB)
  Data is not yet available, as it's currently being analyzed.
Time Frame: 21 days
Measure: Number; unit: mg/m2
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Number analyzed (Participants) | 14
mg/m2
  Cisplatin | 20
  Vinblastine | 1.2
  Temozolomide | 150

3. Primary Outcome: Overall Survival (Phase II)
Description: Overall response rate (complete [CR] or partial response [PR]) according to RECIST version 1.1
Time Frame: Up to 2 years
Measure: Number; unit: participants
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Number analyzed (Participants) | 14
participants
  Partial Response | 3
  Stable Disease | 5
  Progression of Disease | 6

4. Primary Outcome: Maximum Tolerated Dose for RO4929097
Description: based on the incidence of dose-limiting toxicity as assessed the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 (Phase IB)
Time Frame: 21 days
Measure: Number; unit: mg/day
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Number analyzed (Participants) | 14
mg/day | 15

5. Secondary Outcome: Participants' Change in Protein Levels
Description: Participants' pre and post-treatment protein levels will be compared
Time Frame: Baseline up to 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Number analyzed (Participants) | 5
Participants
  decrease in post-treatment cleaved notch protein | 4
  no change | 1

6. Secondary Outcome: Cycle 1 AUC/Pharmacokinetics of Gamma-secretase Inhibitor RO4929097 in Combination With Temozolomide (Phase IB)
Time Frame: Days 4 and 5
Measure: Mean (Standard Deviation); unit: hr·ng/mL
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Number analyzed (Participants) | 5
hr·ng/mL | 5410 (3355)

7. Secondary Outcome: Cycle 1 C Max/Pharmacokinetics of Gamma-secretase Inhibitor RO4929097 in Combination With Temozolomide (Phase IB)
Time Frame: At Cycle 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Number analyzed (Participants) | 5
ng/mL | 301 (172)

8. Secondary Outcome: Cycle 1 Mean Day 2 Trough/Pharmacokinetics of Gamma-secretase Inhibitor RO4929097 in Combination With Temozolomide (Phase IB)
Time Frame: At Day 2 of Cycle 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Number analyzed (Participants) | 5
ng/mL | 129 (88)

9. Secondary Outcome: Number of Participants With Presence or Absence of Markers of Notch Signalling Pathway Inhibition in Patient Tumors (Phase Ib)
Description: The association of response or clinical benefit with the presence or absence of markers of pathway inhibition in patient tumors will be tested using Fisher's exact test.
Time Frame: 2 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Number analyzed (Participants) | 5
Participants
  Insufficient tissue to asses any change | 1
  Sig decrease in post-treatment cleaved Notch | 4

10. Secondary Outcome: Progression-free Survival (Phase II)
Description: Progression-free survival curves will be generated using Kaplan-Meier methodology.
Time Frame: Time from start of treatment to time of progression or death, whichever occurs first, assessed up to 2 years
Measure: Median (Full Range); unit: months
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Number analyzed (Participants) | 14
months | 2.7 [1.2 to 4.1]

11. Secondary Outcome: Participants Evaluated for Toxicity
Description: Number of patients with AE's as assessed by NCI CTCAE v. 4.0 Please see Adverse Events section for specifics.
Time Frame: Up to 30 days post-treatment
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Number analyzed (Participants) | 14
Participants | 14

ADVERSE EVENTS:
Arm/Group | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide)
Serious Adverse Events (participants affected / at risk) | 11/14
Other Adverse Events (participants affected / at risk) | 13/14
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide) (N=14)
Acute kidney injury (Renal and urinary disorders) | 1
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 1
Anemia (Blood and lymphatic system disorders) | 1
Creatinine increased (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 2
Infections and infestations (Infections and infestations) | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 4
Neutrophil count decreased (Blood and lymphatic system disorders) | 5
Pain (General disorders) | 1
Spinal fracture (Musculoskeletal and connective tissue disorders) | 1
White blood cell decreased (Blood and lymphatic system disorders) | 4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (RO4929097, Cisplatin, Vinblastine, Temozolomide) (N=14)
Alanine aminotransferase increased (Blood and lymphatic system disorders) | 4
Alkaline phosphatase increased (Metabolism and nutrition disorders) | 2
Anemia (Blood and lymphatic system disorders) | 11
Anorexia (General disorders) | 1
Aspartate aminotransferase increased (Blood and lymphatic system disorders) | 2
Blood bilirubin increased (Metabolism and nutrition disorders) | 2
CPK increased (Blood and lymphatic system disorders) | 1
Constipation (Gastrointestinal disorders) | 1
Creatinine increased (Metabolism and nutrition disorders) | 4
Diarrhea (Gastrointestinal disorders) | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 1
Fatigue (General disorders) | 4
Flank pain (General disorders) | 2
Hypercalcemia (Metabolism and nutrition disorders) | 1
Hyperglycemia (Metabolism and nutrition disorders) | 12
Hyperkalemia (Metabolism and nutrition disorders) | 4
Hypermagnesemia (Metabolism and nutrition disorders) | 1
Hypertension (Cardiac disorders) | 1
Hypoalbuminemia (Metabolism and nutrition disorders) | 9
Hypocalcemia (Metabolism and nutrition disorders) | 11
Hypoglycemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 4
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 6
Hypophosphatemia (Metabolism and nutrition disorders) | 12
Lipase increased (Metabolism and nutrition disorders) | 1
Lymphocyte count decreased (Blood and lymphatic system disorders) | 10
Nausea (General disorders) | 2
Neck pain (General disorders) | 1
Neutrophil count decreased (Blood and lymphatic system disorders) | 7
Peripheral sensory neuropathy (Nervous system disorders) | 2
Platelet count decreased (Blood and lymphatic system disorders) | 6
Pruritus (Skin and subcutaneous tissue disorders) | 1
Serum amylase increased (Blood and lymphatic system disorders) | 1
Thromboembolic event (Cardiac disorders) | 1
Urinary tract infection (Renal and urinary disorders) | 2
White blood cell decreased (Blood and lymphatic system disorders) | 9

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less